CLINICAL TRIAL: NCT06251687
Title: Application of Transbronchial Cryobiopsy in the Diagnosis of Progressive Pulmonary Fibrosis：a Multicenter Prospective Study
Brief Title: Application of Transbronchial Cryobiopsy in the Diagnosis of Progressive Pulmonary Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZRJY2021-BJ08-03-01-02
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Fibrosis; Transbronchial Cryobiopsy
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transbronchial Cryobiopsy (TBLC) (Experimental): Transbronchial lung cryobiopsy (TBLC) has been increasingly utilised to diagnose diffuse parenchymal lung diseases
  Interventions: Procedure: Transbronchial Cryobiopsy，TBLC
- Transbronchial Lung Biopsy (TBLB) (Active Comparator): Transbronchial lung biopsy (TBLB) is a relatively safe technique routinely employed by pulmonologists for the diagnosis of diffuse parenchymal lung disease
  Interventions: Procedure: Transbronchial Lung Biopsy，TBLB

INTERVENTIONS:
Procedure: Transbronchial Cryobiopsy，TBLC — Transbronchial lung cryobiopsy (TBLC) is a novel technique that has proved its diagnostic value in various diffuse parenchymal lung diseases
  Arms: Transbronchial Cryobiopsy (TBLC)
Procedure: Transbronchial Lung Biopsy，TBLB — Transbronchial lung biopsy (TBLB) is a relatively safe technique routinely employed by pulmonologists for the diagnosis of diffuse parenchymal lung disease
  Arms: Transbronchial Lung Biopsy (TBLB)

SUMMARY:
The goal of this clinical study is to learn about the diagnostic effectiveness, safety, and influencing factors of transbronchial cryobiopsy（TBLC）in progressive pulmonary fibrosis. The main question it aims to answer are: • Determine the prognosis, health economics, and therapeutic strategy changes of patients with TBLC retrograde malleable pulmonary fibrosis. Participants will be randomly divided into two groups, and received TBLB or TBLC.

ELIGIBILITY:
Inclusion Criteria:

Patients with PPF, ≥18 years of age, unclassified ILD, HRCT ≤3 months, forced vital capacity (FVC)≥50% predicted value, pulmonary carbon monoxide diffusion (DLCO)≥35% predicted value, echocardiography ≤12 months, estimated pulmonary systolic blood pressure ≤40 mmHg, Body mass index (BMI)≤35 kg/m2.

Exclusion Criteria:

Patients with platelet counts below 50,000×109/L or International Normalized ratio of prothrombin time (INR) above 1.5 are not eligible for TBLC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the diagnostic performance of transbronchial cryobiopsy（TBLC） | 1 month after transbronchial cryobiopsy
  the sensitivity and specificity of transbronchial cryobiopsy（TBLC）in suspected progressive pulmonary fibrosis

SECONDARY OUTCOMES:
the safety of transbronchial cryobiopsy（TBLC) | 7 days and 1 month after transbronchial cryobiopsy
  The occurence of short-term procedure-related complications, including Bleeding, pneumothorax, death, etc

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China